CLINICAL TRIAL: NCT05626920
Title: A Cross-over Randomized Control Trial to Evaluate the Retinaldehyde Dehydrogenase Inhibitor, Disulfiram, in Improving Retinal Sensitivity in Eyes Affected by Inherited Retinal Degeneration
Brief Title: Disulfiram for Treatment of Retinal Degeneration
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Debarshi Mustafi, Assistant Professor: Dept of Ophthamology, University of Washington
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY00015434
Record Dates: First submitted 2022-11-15; First posted 2022-11-25 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Inherited Retinal Dystrophy Primarily Involving Sensory Retina
MeSH Terms: interventions — Disulfiram

STUDY DESIGN:
Intervention Model Description: Randomized Cross-over study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo medication
  Interventions: Drug: Placebo
- Disulfiram (Active Comparator): Disulfiram medication
  Interventions: Drug: Disulfiram 250 mg

INTERVENTIONS:
Drug: Disulfiram 250 mg — Disulfiram treatment
  Arms: Disulfiram
Drug: Placebo — Placebo treatment
  Arms: Placebo

SUMMARY:
Aberrant retinoic acid signaling driven by the degenerating outer retina leads to pathological changes to the inner retina. The resulting hyperactivity of retinal ganglion cells leads to further diminution of the remaining vision in those afflicted with inherited retinal diseases. Inhibition of this pathway has led to improved visual function in murine models of retinal degeneration. This can be accomplished in humans with the FDA-approved irreversible inhibitor of aldehyde dehydrogenases, disulfiram.

ELIGIBILITY:
Inclusion Criteria:

Age ≥18 years Only those with a clinical diagnosis of inherited retinal degeneration. When available, supporting genetic diagnosis form a CLIA approved lab will be further considered for inclusion.

Only one eye per subject should be identified as the study eye. The study eye must meet the following criteria:

* Best corrected ETDRS visual acuity letter score ≥ 70 (i.e., 20/40 or better) within 30 days of enrollment.
* Goldmann visual field exhibiting constriction of visual fields to 10 degrees centrally
* Able and willing to provide informed consent
* Willing and able to abstain from alcohol consumption for the duration of the study and the 2 weeks preceding it and 2 weeks following the study end point

Liver function values that fall in the normal range as specified below:

* Alanine transaminase (ALT): less than 40 IU/L
* Aspartate transaminase (AST): less than 40 IU/L
* Alkaline phosphatase (ALP): less than 300 IU/L
* Albumin (Alb): less than 50 g/L
* Total Protein: less than 80 g/L
* Total Bilirubin: less than 30 umol/L

Exclusion Criteria:

* A condition that, in the opinion of the investigator, would preclude participation in the study, e.g., alcohol dependence, cardiovascular disease, hepatitis.
* Individuals with a history of diabetes mellitus
* Individuals with a history of psychosis
* Individuals with hypothyroidism
* Individuals with hypersensitivity to thiuram derivatives causing rubber contact dermatitis
* Those on anticoagulant therapy or other medications that may be affected by disulfiram.
* An ocular condition, other than inherited retinal degeneration, is present such that, in the opinion of the investigator, visual acuity might be affected (e.g., foveal atrophy, pigment abnormalities, dense subfoveal hard exudates, non-retinal conditions such as epiretinal membrane or vitreo-macular traction, vein occlusion, uveitis or other ocular inflammatory diseases such as neovascular glaucoma, etc).
* History of major ocular surgery within the prior 6 months or major ocular surgery anticipated within the next 6 months following randomization.
* Exam evidence of severe external ocular infection, including conjunctivitis, chalazion, or substantial blepharitis
* Participation in an investigational trial that involves treatment with any drug within 30 days of randomization that has not received regulatory approval at the time of study entry.

Note: study participants cannot receive another investigational drug while participating in this study.

* Known allergy or hypersensitivity to any component of the study drug.
* For women of child-bearing potential: pregnant or lactating or intending to become pregnant within the next 12 months. Women who are potential study participants should be questioned about the potential for pregnancy. Investigator judgment will be used to determine when a pregnancy test is needed.
* Participants who expect to move out of the area of the clinical center during the 8 months of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-01-03 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Assess the effects of disulfiram on retinal sensitivity in eyes afflicted with inherited retinal degenerations | Year 1
  Evaluate change in contrast sensitivity measured by spatial contrast contrast sensitivity testing between disulfiram and placebo arms

SECONDARY OUTCOMES:
Assess the effects of disulfiram on visual acuity in eyes afflicted with inherited retinal degenerations. | Year 1
  Evaluate change in best corrected visual acuity assessed by ETDRS chart testing between disulfiram and placebo arms
Assess the effects of disulfiram on photoreceptor functionality in eyes afflicted with inherited retinal degenerations. | Year 1
  Evaluate the change in retinal sensitivity as measured by standard and adaptive optics-scanning laser ophthalmoscopy based microperimetry

CONTACTS AND LOCATIONS:
Overall Officials: Debarshi Mustafi, MD, PhD, Principal Investigator — University of Washington
Locations (1):
- University of Washington-South Lake Union Retina Center, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No